CLINICAL TRIAL: NCT01395914
Title: Anamorelin HCl in the Treatment of Non-Small Cell Lung Cancer-Cachexia (NSCLC-C): An Extension Study
Brief Title: Anamorelin HCl in the Treatment of Non-Small Cell Lung Cancer-Cachexia (NSCLC-C): An Extension Study (ROMANA 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-ANAM-303
Record Dates: First submitted 2011-06-30; First posted 2011-07-18 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Cachexia; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Cachexia; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mg QD (Experimental): 100 mg yellow coated, oval tablet; oral administration once daily
  Interventions: Drug: Anamorelin HCl
- Placebo (Placebo Comparator): Placebo tablets identical in appearance to active tablets; oral administration once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anamorelin HCl
  Arms: 100 mg QD
Drug: Placebo
  Arms: Placebo

SUMMARY:
The administration of Anamorelin HCl in patients with Non-Small Cell Lung Cancer-Cachexia (NSCLC-C) is expected to increase appetite, lean body mass, weight gain, and muscle strength.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, placebo-controlled, extension study to assess the safety and efficacy of Anamorelin HCl in NSCLC-C patients.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the Day 85 Visit in the original trial (Study HT-ANAM-301 or HT-ANAM-302) and is considered appropriate to continue to receive additional study drug; must start dosing on the extension study within 5 days of completing dosing on the original trial
* ECOG performance status ≤2
* Life expectancy of >4 months at time of screening
* If woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 30 days following the last dose of study drug (an effective form of contraception is abstinence, a hormonal contraceptive, or a double-barrier method)
* Must be willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Had major surgery (central venous access placement and tumor biopsies are not considered major surgery) within 4 weeks prior to enrollment into the extension study; patients must be well recovered from acute effects of surgery prior to screening; patients should not have plans to undergo major surgical procedures during the treatment period
* Currently taking prescription medications intended to increase appetite or treat weight loss; these include, but are not limited to, testosterone, androgenic compounds, megestrol acetate, methylphenidate, and dronabinol
* Inability to readily swallow oral tablets; patients with severe gastrointestinal disease (including esophagitis, gastritis, malabsorption, or obstructive symptoms) or intractable or frequent vomiting are excluded
* Has an active, uncontrolled infection
* Has known or symptomatic brain metastases
* Receiving strong CYP3A4 inhibitors
* Receiving tube feedings or parenteral nutrition (either total or partial); patients must have discontinued these treatments for at least 6 weeks prior to Day 1, and throughout the study duration
* Other clinical diagnosis, ongoing or intercurrent illness that in the Investigator's opinion would prevent the patient's participation
* Patients actively receiving a concurrent investigational agent, other than Anamorelin HCl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (19):
  - Corona, California
  - Fountain Valley, California
  - Fullerton, California
  - Glendale, California
  - La Jolla, California
  - Riverside, California
  - Washington D.C., District of Columbia
  - Orange City, Florida
  - Quincy, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Lake Success, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Sylvania, Ohio
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Falls Church, Virginia
- Australia (4):
  - Prairiewood, New South Wales
  - Adelaide
  - East Bentleigh
  - Victoria
- Belarus (3):
  - Brest
  - Lesnoy
  - Minsk
- Belgium (5):
  - Antwerp
  - Brussels
  - Genk
  - Ghent
  - Liège
- Canada (4):
  - Edmonton, Alberta
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (5):
  - Benešov
  - Brno
  - Hlučín
  - Liberec
  - Nymburk
- France (2):
  - Lyon
  - Villejuif
- Germany (2):
  - Großhansdorf
  - Halle
- Hungary (2):
  - Budapest
  - Kassai
- Israel (4):
  - Beersheba
  - Petach Tikvah
  - Tel Litwinsky
  - Ẕerifin
- Piacenza, Italy
- Poland (8):
  - Bydgoszcz
  - Grudziądz
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
- Russia (4):
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Yekaterinburg
- Serbia (2):
  - Belgrade
  - Kamenitz
- Ljubljana, Slovenia
- Spain (3):
  - Barcelona
  - Seville
  - Valencia
- Ukraine (3):
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv

REFERENCES:
- [Derived] Currow D, Temel JS, Abernethy A, Milanowski J, Friend J, Fearon KC. ROMANA 3: a phase 3 safety extension study of anamorelin in advanced non-small-cell lung cancer (NSCLC) patients with cachexia. Ann Oncol. 2017 Aug 1;28(8):1949-1956. doi: 10.1093/annonc/mdx192. PMID 28472437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed dosing in either of the original trials of anamorelin HCl in the treatment of NSCLC-C (HT-ANAM-301 or HT-ANAM-302) were able to enroll in this study and continue to receive the study drug to which they were assigned, either anamorelin HCl 100 mg or placebo QD for an additional 12 weeks.
Pre-assignment Details: The primary purpose of this extension study was to permit patients who completed dosing in the original 12-week trials to have the option of continuing to receive randomized study drug for an additional 12 weeks, to further evaluate the safety and tolerability of anamorelin HCl.
Groups:
- Anamorelin HCl: Active drug; 100 mg tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
- Placebo: Placebo tablets identical in appearance to active tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
Period: Overall Study
Arm/Group | Anamorelin HCl | Placebo
Started | 345 | 168
ITT Population | 345 | 168
Safety Population | 343 | 167
Completed | 273 | 131
Not Completed | 72 | 37
Not completed — Unrelated to study drug AE | 6 | 1
Not completed — Death | 23 | 17
Not completed — Other | 9 | 3
Not completed — Withdrawal by patient | 27 | 14
Not completed — Study drug-related AE | 1 | 0
Not completed — Lost to Follow-up | 6 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) Population included all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anamorelin HCl | Placebo | Total
Number analyzed (Participants) | 345 | 168 | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 236 | 120 | 356
  >=65 years | 109 | 48 | 157
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 43 | 126
  Male | 262 | 125 | 387
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 344 | 166 | 510
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Poland | 107 | 60 | 167
  Slovenia | 0 | 1 | 1
  Spain | 5 | 2 | 7
  Belgium | 2 | 2 | 4
  Czech Republic | 11 | 3 | 14
  France | 1 | 2 | 3
  Germany | 3 | 0 | 3
  Hungary | 39 | 16 | 55
  Italy | 1 | 0 | 1
  Netherlands | 1 | 0 | 1
  Canada | 3 | 1 | 4
  United States | 16 | 4 | 20
  Belarus | 8 | 6 | 14
  Israel | 4 | 2 | 6
  Serbia | 4 | 2 | 6
  Ukraine | 64 | 33 | 97
  Russian Federation | 69 | 31 | 100
  Australia | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events
Description: To Evaluate the Safety and Tolerability of Anamorelin HCl.
Time Frame: Over the 12-week treatment period
Population: Safety Population, defined as patients who received any extension trial study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 343 | 167
percentage of participants | 52 | 56

2. Secondary Outcome: Change in Body Weight
Time Frame: Change in body weight from baseline of the original trial through Week 12 of this extension trial.
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 345 | 168
kg | 3.06 (0.631) | 0.92 (0.697)

3. Secondary Outcome: Change in Handgrip Strength of the Non-Dominant Hand
Time Frame: Change in HGS from baseline of the original trial through Week 12 of this extension trial.
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 345 | 168
kg | -0.83 (0.929) | -0.55 (1.036)

4. Secondary Outcome: Change in A/CS Domain Score
Description: Change in the Functional Assessment of Anorexia/Cachexia Treatment (FAACT) 12-item Additional Concerns Subscale (A/CS) domain score is a 12-item scale. Each item is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
  The 12-items are summed together to obtain the domain score. Note that negatively phrased questions are reverse scored so that higher scores always represent improvement/less symptom burden. The total possible score for the A/CS domain ranges from 0 (worst) to 48 (best).
Time Frame: Change in FAACT A/CS Domain Score from baseline of the original trial through Week 12 of this extension trial
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 345 | 168
scores on a scale | 4.46 (0.92) | 3.24 (1.01)

ADVERSE EVENTS:
Time Frame: Adverse events that occurred during the clinical trial, commenced with the first dose of study drug through the 28 day post-treatment follow-up visit.
Description: Adverse events that occurred following the signature of the informed consent, but prior to the first dose of study drug were not reported as adverse events in this trial. The adverse event reporting period also ended if the patient began an alternative therapy within 28 days of the last administration of study drug.
Arm/Group | Anamorelin HCl | Placebo
Serious Adverse Events (participants affected / at risk) | 44/343 | 21/167
Other Adverse Events (participants affected / at risk) | 94/343 | 57/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin HCl (N=343) | Placebo (N=167)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (16) | 7 (7)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (2)
Death (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin HCl (N=343) | Placebo (N=167)
Anaemia (Blood and lymphatic system disorders) | 45 (56) | 25 (37)
Neutropenia (Blood and lymphatic system disorders) | 18 (21) | 8 (8)
Asthenia (General disorders) | 19 (20) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor intends to publish the complete study results in a timely manner that is appropriate to the project. Separate publication of a portion of the study results by any PI is discouraged.